CLINICAL TRIAL: NCT03623126
Title: Impact of ESSURE Devices Withdrawal on the Symptomatology of Patients
Acronym: ESSURE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0160
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Quality of Life; Contraceptive Device; Complications
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — A questionnaire to evaluate clinical improvement and quality of life after ESSURE removal will be completed by patients at least one month after the procedure.

SUMMARY:
The ESSURE device is a method of permanent contraception, marketed in France since 2005. Multiple side effects have been reported by patients since 2015 and the marketing was stopped in 2017. For several months it was observed an increase in requests for withdrawal of these devices. The principal objective of this study is to evaluate clinical improvement and quality of life after ESSURE removal.

This is a multicenter retrospective descriptive study involving the gynecology department of the Croix Rousse Hospital and the gynecology department of the Lyon Sud Hospital over a period of 1 year (1 January 2017-31 December 2017).

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent ESSURE removal due to suspected adverse effects of the device.
* Women who agreed to participate in the study

Exclusion Criteria:

- Women who underwent ESSURE removal to restore their fertility.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women who underwent ESSURE removal between January 2017 and January 2018 in the gynecology department of the Croix Rousse Hospital and the gynecology department of the Lyon Sud Hospital. .
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the clinical improvement after the intervention of withdrawal of ESSURE devices | One day at least one month after the procedure
  This evaluation will be carried out thanks to a questionnaire. The 4th question retrospectively identifies the symptoms presented by patients. The proposed list of symptoms was established by reviewing the symptoms most often found in the medical records of the patients included.
  Question 11 evaluates the variation of each symptom after removal of ESSURE devices through an ordinal scale (total disappearance, significant improvement, poor improvement, no improvement, worsening).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service de gynécologie-Obstétrique - Hôpital de la Croix Rousse, Lyon
  - Service de Gynécologie-Obstétrique - Centre Hospitalier Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No